CLINICAL TRIAL: NCT04348149
Title: Adjunctive Administration of Lindera Obtusiloba on Non-small Cell Lung Cancer Patients Who Receive PD-1 Inhibitors: a Randomized Exploratory Pilot Study
Brief Title: Lindera Obtusiloba for Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun-Yong Choi (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Sponsor-Investigator, Jun-Yong Choi, Professor, Korean Medicine Hospital of Pusan National University
Organization: Korean Medicine Hospital of Pusan National University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PNUKHIRB-2018012
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Dietary Supplement: Lindera obtusiloba extract
- Wait-list (No Intervention)

INTERVENTIONS:
Dietary Supplement: Lindera obtusiloba extract — One package of dietary supplement contains one gram of 70% ethanol extracted powder of Lindera obtusiloba and one gram of glucose powder. Participants intake one package per day for 8 weeks.
  Arms: Intervention group

SUMMARY:
This randomized, open labelled, non-treatment-controlled study evaluates the safety and efficacy of Lindera obtusiloba, a dietary food, on quality of life of non-small cell lung cancer patients who are receiving PD-1 or PD-L1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 20 years
* Patients who have understood and signed the informed consent.
* Subjects who have been confirmed histologically and radiologically for non small cell lung cancer and are scheduled to receive treatment with immune checkpoint inhibitors
* Subjects whose urine HCG are negative and who have agreed with the appropriate method of contraception in case of women of childbearing potential
* Subjects who can fully communicate with their medical doctor about their symptoms or quality of life and who can fill out questionnaires
* Subjects who can follow up during the clinical trial
* Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2
* Hemoglobin ≥ 9g/dL

Exclusion Criteria:

* Subjects who are pregnant, breastfeeding, planning to become pregnant or women of childbearing potential who do not agree with the appropriate method of contraception
* Subjects who have symptomatic and uncontrolled brain or central nervous system metastasis
* Subjects who complain of uncontrolled pain despite using analgesics
* Diastolic Blood Pressure>100mmHg or Systolic Blood Pressure>160mmHg
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels higher than 2.5 times the upper limit for normal
* Creatinine level higher than 1.5 times the upper limit for normal
* Subjects who have participated in other clinical trials within 1 months
* Subjects with a history of serious drug allergies or who have hypersensitivity to the Investigational Product (the main ingredient and its components)
* Subjects with autoimmune diseases
* Subjects who have alcoholism or drug dependence
* Subjects who have cognitive impairment or psychiatric problems
* Subjects who have undergone surgery within 2 weeks
* Subjects who took other herbal medicine or other medicines within 4 weeks
* Subjects who have a medical condition that is likely to affect results or who are determined to be inappropriate to participate in this clinical trial at the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2020-12-27 (Estimated); Study Completion 2020-12-27 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 | Change from baseline to 6-week and 8-week
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30)
EORTC QLQ-LC13 | Change from baseline to 6-week and 8-week
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13)

SECONDARY OUTCOMES:
NK cell percentage in peripheral blood | Change from baseline to 8-week
CD4+/CD8+ T cell in peripheral blood | Change from baseline to 8-week
total T cell, T-helper cell, T-suppressor cell and B-cell percentage in peripheral blood | Change from baseline to 8-week

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Yong Choi, KMD/PHD, Principal Investigator — Korean Medicine Hospital of Pusan National University
Locations (1):
- Korean Medicine Hospital, Pusan National University, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No